CLINICAL TRIAL: NCT01702519
Title: A Pharmacokinetic Evaluation of Two Nicotine Patches in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: RH01418
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-02

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Nicotine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Active Comparator): nicotine transdermal patch with the existing polyisobutylene adhesive
  Interventions: Drug: nicotine
- Treatement (Active Comparator): nicotine transdermal patch with the alternate polyisobutylene adhesive
  Interventions: Drug: nicotine

INTERVENTIONS:
Drug: nicotine — nicotine transdermal patch

SUMMARY:
Bioequivalence study to confirm that a NTS with a polyisobutylene (PIB) adhesive from an alternative supplier delivers the same nicotine blood profile as that of the currently approved NTS with a polyisobutylene adhesive from the current supplier.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-27 kg/m2
* smokes >10 cigarettes per day for preceeding 6 months

Exclusion Criteria:

* inability to stop smoking during study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Celerion NEBRASKA, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single clinical site in the US.
Pre-assignment Details: A total of 128 participants were screened, of which only 40 were randomized into the study. 71 participants did not meet the study eligibility criteria, 4 were lost to follow up, 6 withdrew consent while the remaining 7 were not randomized due to the other reason.
Groups:
- Test Then Reference Patch: Participants first applied a test nicotine patch (21 mg) containing test adhesive for 24 hours, and then entered a washout period of 48 hours. Post-washout, they applied reference nicotine patch containing Reference adhesive (21 mg) for additional 24 hours.
- Reference Then Test Patch: Participants first applied the Reference nicotine patch (21 mg) containing test adhesive for 24 hours, and then entered a washout period of 48 hours. Post-washout, they applied the Test nicotine patch containing reference adhesive (21 mg) for additional 24 hours.
Period: Period 1
Arm/Group | Test Then Reference Patch | Reference Then Test Patch
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Test Then Reference Patch | Reference Then Test Patch
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 2
Arm/Group | Test Then Reference Patch | Reference Then Test Patch
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Then Reference Patch | Reference Then Test Patch | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (11.33) | 31.4 (11.59) | 33.8 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to the Last Quantifiable Sample, AUC(0-t)
Description: Following randomization, the nicotine patches; reference nicotine patch or test nicotine patch (as per the assigned sequence), were applied on participant's upper back or arm. Area under the plasma concentration time curve from zero and extrapolated to the time of last quantifiable sample was determined by plasma concentration time profile of nicotine. Blood samples were drawn at the following time intervals: immediately pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 20, 24, 25, 26, 28, and 32 hours after the application of the patch. Patch was then removed after the collection of 24 hour blood sample. AUC(0 -t) was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: Baseline to 32 hours
Population: Per Protocol Population, which consisted of all randomized participants who took at least one dose of the study treatment, did not have any protocol deviation, and provided enough pharmacokinetic data as determined by the pharmacokineticist.
Measure: Mean (Standard Deviation); unit: nanogram (ng)*hour (hr)/milliliter (mL)
Groups:
- Test Patch: Participants were instructed to wear transdermal nicotine patch (21 mg) with test adhesive, for 24 hours.
- Reference Patch: Participants were instructed to wear transdermal nicotine patch (21 mg) with the reference adhesive, for 24 hours.
Arm/Group | Test Patch | Reference Patch
Number analyzed (Participants) | 38 | 38
nanogram (ng)*hour (hr)/milliliter (mL) | 494.54 (115.075) [0.92 to 1.0] | 528.43 (129.762) [0.91 to 0.98]
Statistical Analysis 1: Comparison: Test Patch vs Reference Patch; Null hypothesis considered no difference between the two treatments; Test type: Non-Inferiority or Equivalence — Bio-equivalence was established if 90% confidence interval (CI) of the ratio (Test/Ref) of geometric means was included in the limit of 0.80 - 1.25; Treatment Ratio; Treatment Ratio = 0.946, 90% CI 2-sided [0.912 to 0.982] — The ratio between the geometric means of the test and reference formulations was calculated

2. Primary Outcome: Maximum Measured Plasma Concentration (Cmax)
Description: Following randomization, the nicotine patches; reference nicotine patch or test nicotine patch (as per the assigned sequence), were applied on participant's upper back or arm. Maximum plasma nicotine concentration was determined from plasma concentration time profiles. Blood samples were drawn at various time points: immediately pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 20, 24, 25, 26, 28, and 32 hours after application the patch. Patch was then removed after the collection of 24 hour blood sample. Cmax was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: Baseline to 32 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Patch | Reference Patch
Number analyzed (Participants) | 38 | 38
ng/mL | 22.31 (4.986) | 23.50 (5.917)
Statistical Analysis 1: Comparison: Test Patch vs Reference Patch; Null hypothesis considered no difference between the treatments; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if 90% confidence interval (CI) of the ratio (Test/Ref) of geometric means was included in the limit of 0.80 - 1.25; Treatment Ratio; Treatment Ratio = 0.962, 90% CI 2-sided [0.92 to 1.00] — The ratio between the geometric means of the test and reference formulations was calculated

3. Secondary Outcome: Area Under the Concentration Time Curve Between Zero and Infinity, AUC (0-inf)
Description: Following randomization, the nicotine patches; reference nicotine patch or test nicotine patch (as per the assigned sequence), were applied on participant's upper back or arm. Area under the plasma nicotine concentration time curve from zero extrapolated to infinity was determined by plasma concentration time profile of nicotine. Blood samples drawn at various time points including: immediately pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 20, 24, 25, 26, 28, and 32 hours after wearing the patch. Patch was then removed after the collection of 24 hour blood sample. AUC(0 -inf) was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: Baseline to 32 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Reference Patch: Participants were instructed to wear transdermal nicotine patch (21 mg) with reference adhesive, for 24 hours
Arm/Group | Test Patch | Reference Patch
Number analyzed (Participants) | 38 | 38
ng*h/mL | 505.13 (118.939) | 541.15 (134.854)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Following randomization, the nicotine patches; reference nicotine patch or test nicotine patch (as per the assigned sequence), were applied on participant's upper back or arm. Time to Maximum Plasma Concentration was determined from plasma concentration time profiles. Blood samples were drawn at various time points; immediately pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 20, 24, 25, 26, 28, and 32 hours after application of the patch. Patch was then removed after the collection of 24 hour blood sample. Tmax was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: Baseline to 32 hours
Population: Per protocol population, which included all randomized participants who took at least one dose of the drug, did not have any protocol deviations and whose data was considered evaluable by the pharmacokineticist.
Measure: Median (Full Range); unit: hrs
Groups:
- Test Patch: Participants were instructed to wear transdermal nicotine patch with test adhesive, for 24 hours.
- Reference Patch: Participants were instructed to wear transdermal nicotine patch with reference adhesive, for 24 hours.
Arm/Group | Test Patch | Reference Patch
Number analyzed (Participants) | 38 | 38
hrs | 10.00 [0.5 to 24.0] | 17.99 [2.0 to 24.0]

5. Secondary Outcome: Plasma Half-life (t1/2)
Description: Following randomization, the nicotine patches; reference nicotine patch or test nicotine patch (as per the assigned sequence), were applied on participant's upper back or arm. The elimination half-life of nicotine was determined by from plasma concentration time profiles. Blood samples were drawn at several time points: immediately pre-dose, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 20, 24, 25, 26, 28, and 32 hours after the application of the patch. Patch was then removed after the collection of 24 hour blood sample. Plasma half-life (t1/2) was based on the baseline adjusted nicotine plasma concentration data
Time Frame: Baseline to 32 hours
Population: Per-prorocol population, which included all randomized participants who received at least one dose of the study treatment, had no protocol violation, and whose data was considered evaluable by the pharmacokineticist.
Measure: Median (Full Range); unit: Hrs
Arm/Group | Test Patch | Reference Patch
Number analyzed (Participants) | 38 | 38
Hrs | 2.55 [2.0 to 3.5] | 2.59 [2.0 to 3.7]

6. Secondary Outcome: Rate of Elimination (Kel)
Description: Following randomization, the nicotine patches; reference nicotine patch or test nicotine patch (as per the assigned sequence), were applied on participant's upper back or arm. Elimination rate constant for nicotine was determined from plasma concentration time profiles. Blood samples were drawn at several time points: immediately pre-dose, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 20, 24, 25, 26, 28, and 32 hours the application of the patch. Patch was then removed after the collection of 24 hour blood sample. Elimination rate constant for nicotine was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: Baseline to 32 hours
Population: Per protocol population, which included all randomized participants who took at least one dose of the study medications, had no protocol violations, and whose data was considered evaluable by the pharmacokineticist.
Measure: Median (Full Range); unit: 1/hr
Arm/Group | Test Patch | Reference Patch
Number analyzed (Participants) | 38 | 38
1/hr | 0.27 [0.2 to 0.3] | 0.27 [0.2 to 0.3]

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of the smoking abstinence sequestration period and until five days following last administration of the study treatments
Arm/Group | Test Patch | Reference Patch
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 22/38 | 26/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Patch (N=38) | Reference Patch (N=39)
Application Site Erythema (General disorders) | 15 (15) | 20 (20)
Application Site Pruritus (General disorders) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.